CLINICAL TRIAL: NCT00256178
Title: A Placebo-controlled, Double-blind, Randomized Study to Evaluate the Efficacy and Safety of TAK-475 50 mg and 100 mg Versus Placebo, When Co-administered With Simvastatin 20 mg or 40 mg in Subjects With Primary Dyslipidemia.
Brief Title: Efficacy of Lapaquistat Acetate and Simvastatin in Subjects With Primary Dyslipidemia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-475/EC302; 2005-002313-21 (EudraCT Number); U1111-1122-8212 (Registry Identifier: WHO)
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Hypercholesterolemia
Keywords: Hyperlipidemia; Drug Therapy
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lapaquistat Acetate 50 mg QD + Simvastatin (Experimental)
  Interventions: Drug: Lapaquistat acetate and simvastatin
- Lapaquistat Acetate 100 mg QD + Simvastatin (Experimental)
  Interventions: Drug: Lapaquistat acetate and simvastatin
- Simvastatin (Active Comparator)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Lapaquistat acetate and simvastatin — Lapaquistat acetate 50 mg, tablets, orally, once daily and stable simvastatin therapy for up to 24 weeks.
  Other Names: Lapaquistat; Zocor; TAK-475
  Arms: Lapaquistat Acetate 50 mg QD + Simvastatin
Drug: Lapaquistat acetate and simvastatin — Lapaquistat acetate 100 mg, tablets, orally, once daily and stable simvastatin therapy for up to 24 weeks.
  Other Names: Lapaquistat; Zocor; TAK-475
  Arms: Lapaquistat Acetate 100 mg QD + Simvastatin
Drug: Simvastatin — Lapaquistat acetate placebo-matching tablets, orally, once daily and stable simvastatin therapy for up to 24 weeks.
  Other Names: Zocor
  Arms: Simvastatin

SUMMARY:
The purpose of the study is to determine the efficacy of lapaquistat acetate, once daily (QD), taken with simvastatin on cholesterol levels in subjects with primary dyslipidemia

DETAILED DESCRIPTION:
In humans, cholesterol is acquired from dietary sources and is produced de novo in the liver, intestine, and various other tissues. Normally, the balance among cholesterol synthesis, dietary intake, and degradation is adequate to maintain healthy cholesterol plasma levels; however, in subjects with hypercholesterolemia, elevation in low-density lipoprotein cholesterol leads to atherosclerotic deposition of cholesterol in the arterial walls (atherosclerosis) and subsequent coronary heart disease. Thus, it has been established that lowering the low-density lipoprotein cholesterol plasma concentrations effectively reduces cardiovascular morbidity and mortality. Additional lipid risk factors for coronary heart disease include elevated triglyceride, very low-density lipoprotein cholesterol and low-density lipoprotein cholesterol levels, and low levels of high-density lipoprotein cholesterol.

Despite changes in lifestyle and the availability of potent lipid-lowering agents, cardiovascular disease continues to be the major cause of death in Western Europe and North America. Serum cholesterol levels exceeding 5 mmol/L (193 mg/dL) are common in adults in Britain and much of Europe, the United States, Australia, and New Zealand, representing a serious public health concern.

Currently, 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitors (ie, statins) are the first-line monotherapies prescribed for the treatment of dyslipidemia, after diet and therapeutic lifestyle changes alone fail to reduce low-density lipoprotein cholesterol to desired levels. Statins reduce low-density lipoprotein cholesterol and triglycerides, increase high-density lipoprotein cholesterol, and improve endothelial function. Treatment with statins reduces the risk of a vascular event by about 30% in subjects with and without symptoms of arteriosclerosis; however, many subjects fail to reach recommended levels of low-density lipoprotein cholesterol reduction after receiving low-dose statins as a monotherapy. Consequently, the dosage of statins is often increased or an additional treatment is added; the latter has become an important therapeutic option for achieving increasingly stringent lipid targets set forth by international therapeutic guidelines.

Simvastatin, a long-established treatment for dyslipidemia as monotherapy or in combination with other drugs, is a lactone that, once hydrolyzed, inhibits 3-hydroxy-3-methylglutaryl coenzyme A reductase. At the molecular level, the rate of synthesis of cholesterol depends primarily on the highly regulated activity of 3-hydroxy-3-methylglutaryl coenzyme A reductase.

TAK-475 (lapaquistat acetate) is a squalene synthase inhibitor currently under development at Takeda for the treatment of dyslipidemia. This study will evaluate the efficacy and safety of lapaquistat acetate taken with simvastatin in subjects with hypercholesterolemia. Total participation time in this study is expected to be up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential who are sexually active must agree to use adequate contraception from screening throughout the duration of the study and for 30 days following the last dose.
* Has a documented history of dyslipidemia with or without cardiovascular risk factors but without type 1 or 2 diabetes.
* Is on a stable dose of simvastatin, either 20 or 40 mg, for at least 4 weeks prior to Screening.
* Prior to Randomization, the participant has a mean low density lipoprotein cholesterol level greater than or equal to 100 mg/dL and less than or equal to 190 mg/dL for 2 consecutive samples.
* Prior to Randomization, the subject has mean triglyceride level greater than or equal to 400 mg/dL for 2 consecutive samples.
* Is willing and able to comply with the recommended, standardized diet.

Exclusion Criteria:

* Has annine aminotransferase or aspartate aminotransferase level greater than 1.5 times the upper limit of normal, identified during screening.
* Has a serum creatinine greater than 133 mmol/L, identified during screening.
* Has a creatine kinase greater than 3 times the upper limit of normal, identified during screening.
* Has active liver disease or jaundice.
* Has taken any bile acid sequestrants [eg, cholestyramine], and intestinal cholesterol uptake inhibitors [eg, ezetimibe]) from 30 days before Screening until study completion or any fibrates for 6 weeks before Visit 1.
* Has a previous history of cancer that has been in remission for less than 5 years prior to the first dose of study medication.
* Has an endocrine disorder, such as Cushing's syndrome, hyperthyroidism, or inappropriately treated hypothyroidism affecting lipid metabolism.
* Has a history of myocardial infarction, angina pectoris, unstable angina, transient ischemic attacks, cerebrovascular accident, peripheral vascular disease, abdominal aortic aneurysm, coronary angioplasty, coronary or peripheral arterial surgery, or multiple risk factors that confer a 10-year risk for cardiovascular heart disease greater than 20% based on Framingham risk scoring.
* Has a positive hepatitis B surface antigen or hepatitis C virus antibody test, as determined by medical history.
* Has a positive human immunodeficiency virus status or is taking antiretroviral medications, as determined by medical history and/or subject's verbal report.
* Has received any investigational medication 30 days prior to screening, (for drugs with a long half-life, within a period of less than 5 times the drug's half-life) or is participating in an investigational study.
* Has received lapaquistat acetate in a previous clinical study or as a therapeutic agent.
* Has a history or presence of clinically significant food allergy that would prevent adherence to the specialized diet.
* Has a known heterozygous or homozygous familial hypercholesterolemia or known type III hyperlipoproteinemia (familial dysbetalipoproteinemia).
* Has fibromyalgia, myopathy, rhabdomyolysis, or unexplained muscle pain.
* Has uncontrolled hypertension
* Has had inflammatory bowel disease or any other malabsorption syndrome, or has had gastric bypass or any other surgical procedure for weight loss.
* Has a history of drug abuse or a history of high alcohol intake within the previous 2 years.
* Has type 1 or 2 diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2005-10; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in fasting plasma Low Density Lipoprotein cholesterol | Week 24 or Final Visit

SECONDARY OUTCOMES:
Change from Baseline in Triglycerides | Week 24 or Final Visit
Change from Baseline in Total Cholesterol | Week 24 or Final Visit
Change from Baseline in High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in Very Low Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in apolipoprotein A1 | Week 24 or Final Visit
Change from Baseline in apolipoprotein B | Week 24 or Final Visit
Change from Baseline in non- High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in the ratio of Low Density Lipoprotein cholesterol/High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in the ratio of Total Cholesterol/High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in the ratio of apolipoprotein A1/apolipoprotein B | Week 24 or Final Visit
Change from Baseline in high-sensitivity C-reactive protein | Week 24 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 1.81 mmol/L (70 mg/dL) | Week 24 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 2.59 mmol/L (100 mg/dL) | Week 24 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 3.37 mmol/L (130 mg/dL) | Week 24 or Final Visit
Best corrected visual acuity | Week 24 or Final Visit
Adverse Events | Weeks 2, 4, 8, 12, 16, 20, and 24 or Final Visit
Clinical Laboratory Tests | Weeks 2, 4, 8, 12, 16, 20, and 24 or Final Visit
Vital Signs | Weeks 2, 4, 8, 12, 16, 20, and 24 or Final Visit
12-lead Electrocardiogram | Timeframe: Weeks 12 and 24 or Final Visit
Physical Examination | Week 24 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (53):
- Czechia (9):
  - Benešov
  - Holice V Čechách
  - Kladno
  - Mladá Boleslav
  - Olomouc
  - Prague
  - Trutnov
  - Ústí nad Orlicí
  - Zlín
- Estonia (3):
  - Pärnu
  - Tallinn
  - Tartu
- Finland (6):
  - Aura
  - Helsinki
  - Hyvinkää
  - Oulu
  - Tampere
  - Turku
- Germany (8):
  - Berlin
  - Bochum
  - Chemnitz
  - Dresden
  - Frankfurt
  - Görlitz
  - Leipzig
  - Nuremberg
- Poland (9):
  - Krakow
  - Lublin
  - Niemodlin
  - Skierniewice
  - Sroda Wlkp.
  - Starachowice
  - Swietokrzyski
  - Warsaw
  - Zakopane
- South Africa (6):
  - Bloemfontein
  - Cape Town
  - Johannesburg
  - Pretoria
  - Randburg
  - Tongaat
- United Kingdom (12):
  - Bath
  - Birmingham
  - Blackpool
  - Blantyre
  - Chippenham
  - Eastwood
  - Glasgow
  - Harrow
  - Hinckley
  - Newport Isle of Wight
  - Nottingham
  - Woolpit

REFERENCES:
- [Result] Stein EA, Bays H, O'Brien D, Pedicano J, Piper E, Spezzi A. Lapaquistat acetate: development of a squalene synthase inhibitor for the treatment of hypercholesterolemia. Circulation. 2011 May 10;123(18):1974-85. doi: 10.1161/CIRCULATIONAHA.110.975284. Epub 2011 Apr 25. PMID 21518985